CLINICAL TRIAL: NCT00994929
Title: Phase II Biologic Effects Study of Recombinant Interleukin-11 (rhIL-11, Neumega) in Subjects With Moderate or Mild Hemophilia A, or Von Willebrand Disease Unable to Use DDAVP
Brief Title: Efficacy and Safety of IL-11 in DDAVP Unresponsive
Acronym: IL-11DDAVP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Margaret Ragni, Laurel Yasko, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO08070154, Wyeth 3067K1-2214
Record Dates: First submitted 2009-10-12; First posted 2009-10-14 (Estimated); Results first posted 2016-03-02 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-02

CONDITIONS: Hemophilia A; Von Willebrand Disease
Keywords: biologic effects; von Willebrand disease; hemophilia; interleukin-11; DDAVp
MeSH Terms: conditions — Hemophilia A; von Willebrand Diseases | interventions — oprelvekin; Interleukin-11

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Neumega (Oprelveken, Interleukin 11) (Experimental): Neumega (Oprelveken, interleukin-11 (IL-11) 25 microgram/kilogram by subcutaneou injection once daily for four days, followed on day 4 DDAVP 0.3 microgram/kilogram intravenously 30 minutes after neumega
  Interventions: Biological: Neumega (Oprelvekin, Interleukin 11, IL-11)

INTERVENTIONS:
Biological: Neumega (Oprelvekin, Interleukin 11, IL-11) — 25 microgram/kg IL-11 by subcutaneous injection once daily for four days, followed by DDAVP 0.3 microgram/kg by intravenous infusion over 30 minutes on day 4, 30 minutes after IL-11.
  Other Names: Interleukin-11; IL-11; Oprelvekin

SUMMARY:
The purpose of this study is to determine the biologic efficacy and safety of rhIL-11 when given subcutaneously in adults with moderate or mild hemophilia A or Von Willebrand disease unresponsive to DDAVP. Biologic efficacy will be measured by the number and percent increase of VWD coagulation tests (FVIII:C, VWF: Ag, VWF: RCo, closure time, APTT, and VWF multimers) to the normal range, or at least to 1.5-3 time baseline, following dosing of rhIL-11 when given daily for 4 days, and boosted by DDAVP infusion on day 4, in those in whom DDAVP is not contraindicated. Safety will be measured by the frequency of adverse events, including fever, headache, fatigue, myalgias, arthralgias, fluid retention, or edema.

DETAILED DESCRIPTION:
This is a prospective, single center, Phase II biologic effects study of recombinant interleukin-11 (rhIL-11, Neumega) in subjects hemophilia A, moderate or mild; or with Von Willebrand disease unable to take desmopressin acetate (DDAVP) because they are unresponsive, allergic, or DDAVP is contraindicated. The purpose of the study is to establish the biologic efficacy and safety of rhIL-11 in those not able to take DDAVP. Study subjects will include adults, age >= 18 years, with hemophilia A, moderate, defined as factor VIII 0.01-0.04 U/ml, or mild, defined as factor VIII >= 0.05 U/ml; or with VWD defined by low VWF:RCo and /or low VWF:Ag, past bleeding history, and/or family history of VWD. A total of 10-16 subjects will be enrolled in order to assure that 10 complete the study. The specific aims of the study are: 1) to determine the biologic effect of rhIL-11 when given 4 consecutive days; 2) to determine the safety of rhIL-11 when used in subjects with hemophilia A, moderate or mild; or with VWD unresponsive or unable to take DDAVP; and 3) to determine the mechanism of the hemostatic effects of rhIL-11. The biologic efficacy outcomes will be measured by VWD-related coagulation tests (VWF:RCo, FVIII:C, VWF:Ag, closure times) before and after rhIL-11 injection. Safety outcomes will be measured by the number and frequency of adverse events, including fever, headache, fatigue, myalgias, arthralgias, fluid retention, or edema. The mechanism of rhIL-11 hemostatic effect will be measured by VWFmRNA before and after rhIL-11 response. Response to DDAVP following rhIL-11 will also be assessed in those in whom DDAVP is not contraindicated. The study will last up to 1 month per subject, and for 24 months for the entire study.

ELIGIBILITY:
Inclusion Criteria:

* Males or females >= 18 years of age.
* A diagnosis of hemophilia A, moderate (FVIII:C 0.01-0.04 U/ml) or mild (FVIII:C >= 0.05 U/ml); or a diagnosis of VWD, defined by a low VWF:RCo and past bleeding history.
* For those with VWD, an inability to use DDAVP due to i) unresponsiveness defined as VWF:RCo or FVIII:C level lower than 50 IU/dl or less than a 3-fold increase after 0.3 microgram/kg DDAVP; ii) allergic reactions or seizures; or iii) a contraindication to DDAVP.
* Willingness to have blood drawn.
* Willingness to sign informed consent.

Exclusion Criteria:

* Presence of other bleeding disorders, acquired Von Willebrand disease, primary thrombocytopenia.
* Use of immunomodulatory or experimental drugs, or diuretics.
* Pregnant or lactating women.
* Previous cardiac disease, congestive failure, arrhythmia (e.g. atrial fibrillation, atrial flutter), hypertension, MI, stroke, or thrombosis.
* Past allergic reaction to Neumega.
* Surgery within the past 8 weeks.
* Inability to comply with study protocol requirements.
* Concomitant use of antiplatelet drugs, anticoagulants, dextran, aspirin or NSAIDs.
* Treatment with DDAVP, cryoprecipitate, whole blood, plasma and plasma derivatives containing substantial quantities of FVIII and/or VWF within five days of study.
* Baseline safety and/or hematology lab values outside the normal limits and/or an EKG indicating an arrhythmia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2010-01; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret V. Ragni, MD, MPH, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Ragni MV, Jankowitz RC, Chapman HL, Merricks EP, Kloos MT, Dillow AM, Nichols TC. A phase II prospective open-label escalating dose trial of recombinant interleukin-11 in mild von Willebrand disease. Haemophilia. 2008 Sep;14(5):968-77. doi: 10.1111/j.1365-2516.2008.01827.x. Epub 2008 Aug 1. PMID 18680527
- [Derived] Ragni MV, Novelli EM, Murshed A, Merricks EP, Kloos MT, Nichols TC. Phase II prospective open-label trial of recombinant interleukin-11 in desmopressin-unresponsive von Willebrand disease and mild or moderate haemophilia A. Thromb Haemost. 2013 Feb;109(2):248-54. doi: 10.1160/TH12-06-0447. Epub 2012 Dec 13. PMID 23238591

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Nine (9) subjects 18 years or older, including five with mild or moderate hemophilia A (HA) and four with mild or moderate von Willebrand disease (VWD) unresponsive or allergic to DDAVP were enrolled in and completed the study between January 2010 and February 2012.
Pre-assignment Details: Following enrollment, subjects initiated study drug.
Groups:
- Neumega (Oprelveken, Interleukin 11): 25 µg/kilogram of body weight of rhIL-11 subcutaneously administered on days 1 to 4. On day 4 following rhIL-11 injection DDAVP was subsequently given at 0.3 mcg/kg intravenously over 30 minutes. For any subject with past allergic reactions, hypersensitivity, or seizures with DDAVP, or in whom DDAVP is contraindicated, DDAVP was not given: only rhIL-11 was given on Day 4.
Period: Overall Study
Arm/Group | Neumega (Oprelveken, Interleukin 11)
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 5 subjects were mild or moderate hemophilia A; 4 were mild or moderate VWD; all unresponsive or allergic to DDAVP The VWD subjects - 2, type 1 and 2, type 2 VWD, including one with type 2B, and one with type 2M. All subjects had positive past bleeding histories.
Groups:
- Neumega (Oprelveken, Interleukin 11): The VWD subjects included two with type 1 VWD and two with type 2 VWD, including one with type 2B, with increased platelet aggregation at low strength ristocetin and absent high molecular weight multimers, and one with type 2M disease, with reduced VWF:RCoF/ VWF:Ag ratio <0.50, per NHLBI criteria (Table 2).5 All subjects had positive past bleeding histories. Pregnancy, lactation, heart disease, uncontrolled hypertension, arrhythmia, thrombosis, recent surgery or receipt of blood products were exclusions. A total of nine subjects were enrolled and completed study, including five with hemophilia A and four with VWD. The median age was 26 years, range 22-51 years
Arm/Group | Neumega (Oprelveken, Interleukin 11)
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 26 [22 to 51]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Biologic Effects by Coagulation Tests
Description: VWF activity was measured by ristocetin-induced platelet agglutination using a Chronolog aggregometer11-14 and VWF:Ag by "sandwich" ELISA, using anti-VWF antibodies (DakoA082, Carpintera CA). Results were expressed in percent, with normal human plasma pool designated 100%, and severe type 3 VWD plasma used as the negative control
Time Frame: within 4 days of study drug.
Population: Four subjects had VWD and five subjects had mild hemophilia A
Measure: Mean (Standard Error); unit: percentage of normal
Arm/Group | Neumega (Oprelveken, Interleukin 11)
Number analyzed (Participants) | 9
percentage of normal
  VWD patients | 34.75 (19.2)
  Mild hemophilia A patients | 143.4 (18.6)

2. Secondary Outcome: The Frequency of Adverse Events
Time Frame: within 11 days of study drug
Measure: Number; unit: participants
Arm/Group | Neumega (Oprelveken, Interleukin 11)
Number analyzed (Participants) | 9
participants | 6

3. Secondary Outcome: The Mechanism of Study Drug Effect by VWF mRNA.
Time Frame: within 11 days of study drug.
Measure: Mean (Full Range); unit: fold increase
Arm/Group | Neumega (Oprelveken, Interleukin 11)
Number analyzed (Participants) | 9
fold increase | 0.81 [-0.07 to 2.65]

ADVERSE EVENTS:
Time Frame: January 2010 to February 2012
Groups:
- Neumega (Oprelveken, Interleukin 11): Neumega (Oprelvekin, Interleukin 11, IL-11): 25 microgram/kg IL-11 by subcutaneous injection once daily for four days, followed on day 4 by DDAVP 0.3 microgram/kg by intravenous infusion.
Arm/Group | Neumega (Oprelveken, Interleukin 11)
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 6/9
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neumega (Oprelveken, Interleukin 11) (N=9)
Conjunctival Infection (Eye disorders) | 6 (6) — Grade 1 or less
Dyspepsia (Gastrointestinal disorders) | 3 (3)
Fluid Retention (General disorders) | 2 (2)
Flu-Like Symptoms (General disorders) | 2 (2)
Headache (General disorders) | 2 (2)
Injection Site Erythema (General disorders) | 2 (2)
Lightheadedness (General disorders) | 1 (1)
Flushing (General disorders) | 1 (1)
Insomnia (General disorders) | 1 (1)
Drowsiness (General disorders) | 1 (1)
Hyponatremia (General disorders) | 1 (1) — Hyponatremia occurred in a diabetic patient after excess fluid intake for symptomatic hyperglycemia, which resolved with fluid restriction. Hyponatremia was grade 3 (129 mEq/L).
Thrombocytopenia (General disorders) | 2 (2) — One of the two patients with thrombocytopenia was the 2B VWD patient, whose baseline platelet count was low and remained unchanged after rhIL-11.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No